CLINICAL TRIAL: NCT05120765
Title: A Pilot Randomized Controlled Trial of The CONNECT Program: Testing a Telephone-Based Mental Health Intervention in a Clinical Sample of Socially Isolated Older Adults
Brief Title: The CONNECT Program: Testing a Telephone-Based Mental Health Intervention for Older Adults
Acronym: CONNECT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in study design was implemented and the study design no longer follows a pilot randomized controlled trial.
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Inga Christianson, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HE2021-0124
Record Dates: First submitted 2021-10-17; First posted 2021-11-15 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Social Isolation; Loneliness; Depression; Anxiety
Keywords: Mental health problems; Adults 65+; Loneliness; Social Isolation; Intervention; Telephone therapy; Group therapy; Aging; Older adults; Clinical; Acceptance and Commitment Therapy; Self-compassion; Mindfulness
MeSH Terms: conditions — Social Isolation; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention to be administered is "The CONNECT Program". This is a 6-week, group-based, telephone-based, mental health intervention for socially isolated older adults. This group-therapy intervention is based on principles of Acceptance and Commitment Therapy (ACT).
  Interventions: Behavioral: The CONNECT Program
- Waitlist (No Intervention): Waitlist intervention requires participants to wait 6 weeks. This waitlist group will receive the intervention after this 6 week waiting period, due to the exploratory nature of this Pilot Randomized Controlled Trial (RCT).

INTERVENTIONS:
Behavioral: The CONNECT Program — The CONNECT Program is a 6-week, group-based, telephone-based, mental health intervention for socially isolated older adults. This group-therapy intervention is based on principles of Acceptance and Commitment Therapy (ACT). The group sessions take place once a week and they last 90 minutes each.
  Arms: Intervention

SUMMARY:
This study will test a telephone-based group intervention called "The CONNECT Program" which is designed for adults aged 65+ who are currently experiencing social isolation or loneliness, and symptoms of anxiety or depression. A pilot randomized controlled trial (RCT) will be conducted to evaluate The CONNECT Program using a clinical sample of adults 65+. The goals of this research include, (a) testing the feasibility of conducting a large-scale RCT using a clinical sample of adults 65+; (b) understanding the experiences of this clinical sample of adults 65+ in The CONNECT Program; and (c) investigating the preliminary effectiveness of this program with this sample. Participants (N=16) will be randomly assigned to either the waitlist or intervention group. Both groups will receive the intervention and share their experiences in The CONNECT Program. The waitlist group will receive the intervention after the waiting period. All participants will complete questionnaires before receiving the intervention, after receiving the intervention, and each week during the intervention. This study will provide us with insight regarding what this clinical sample of participants think of The CONNECT Program, how we can improve the program in the future in order to meet the needs of this group, what changes to the study design are needed in order to execute a large-scale randomized controlled trial in the future, and if this program shows preliminary effectiveness in this sample.

DETAILED DESCRIPTION:
The population of adults aged 65+ in Canada is increasing (Statistics Canada, 2019). Some of the most common mental health and psychosocial problems experienced by adults aged 65+ include anxiety, depression, social isolation, and loneliness. The current research will test a telephone-based group intervention called "CONNECT" which is designed for adults aged 65+ who are currently experiencing social isolation or loneliness, and symptoms of anxiety or depression. CONNECT stands for: "Creating Opportunities to build social Networks, learn New skills to manage challenging emotions Enhance mindful awareness and acceptance of emotions, and increase self-Compassion, through Telephone-based group programming". A pilot randomized controlled trial will be conducted to evaluate The CONNECT Program using a clinical sample of adults 65+ recruited from Winnipeg and Brandon.

We will use a randomized design to pilot this intervention and assess the feasibility of implementing and testing this intervention with a clinical sample of adults 65+. Participants will be randomized 1:1 to one of two conditions (1 = intervention, 2 = waitlist). The quantitative data we collect will inform us about changes in self-reported symptoms on the primary and secondary outcome measures and it will reveal information about treatment satisfaction and how participants experienced each session. Additionally, the questionnaire that will be administered after each session and the post-CONNECT questionnaire will include open-ended questions where participants can expand on their answers about treatment satisfaction and their experiences in the program.

Within one week before the first CONNECT session, all participants will complete the baseline questionnaire and will then be randomized to one of two groups (1 = intervention, 2 = waitlist). One week after the baseline questionnaire is complete, participants in the intervention group will receive six weeks of CONNECT group therapy, and participants in the waitlist group will begin the waiting period. Within one week of the last CONNECT session, all participants will complete the post-CONNECT questionnaire. Participants receiving the intervention will also complete the Group Session Rating Scale (GSRS) after each session in order to monitor the participant progress from session to session and to evaluate the group-therapy alliance. Due to the exploratory nature of this pilot RCT, participants in the waitlist group will complete the baseline questionnaire again, they will receive the intervention and complete the GSRS each week, and they will complete post-CONNECT questionnaire one week after the last session. We plan to collect this data because we want to capture the experiences of the waitlist participants both when they are waiting for the intervention and when they receive the intervention. The purpose of including a waitlist group is to help determine if the current study procedures are acceptable. This will allow us to better understand potential issues such as participant dropout, and it will help us identify changes that should be made for a future RCT.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older, currently living in Manitoba, self-reporting symptoms of social isolation and/or loneliness, and self-reporting symptoms of depression and/or anxiety.

Exclusion Criteria:

* Under 65 years of age, living outside of Manitoba, being unable to provide consent independently, deafness not corrected by hearing aids (hearing is needed as this is a telephone program), an absence of self-reported symptoms of anxiety or depression, an absence of symptoms of loneliness or social isolation, self-reporting suicidal ideation or suicidal behaviours that are current, substance use or substance dependence within the past six months, bipolar I or II, psychotic disorders, and major neurocognitive disorders. Another exclusion criteria would be an individual who does not have access to a telephone, or is not comfortable using the telephone for the purpose of The CONNECT Program or The research components (i.e., the questionnaires).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Treatment Satisfaction and Feedback | Immediately after session 1, immediately after session 2, immediately after session 3, immediately after session 4, immediately after session 5, immediately after session 6, immediately after the intervention ends
  Measured using Group Session Rating Scale (Duncan & Miller, 2007), and open-ended questions in the post-CONNECT questionnaire. Reference: Duncan, B., & Miller, S. (2007). The Group Session Rating Scale. Jensen Beach, FL: Author.
Acceptance and Action Questionnaire II (AAQ-II) (Bond et al., 2011). | 1 week before the intervention begins, immediately after intervention ends (approximately 7 weeks)
  Measures psychological flexibility
PROMIS (Patient-Reported Outcomes Measurement Information System) Depression Short Form 4a (Cella et al., 2010; Cella et al., 2019) | 1 week before the intervention begins, immediately after intervention ends (approximately 7 weeks)
  Measures symptoms of depression
The PROMIS Anxiety Short Form 4a (Cella et al., 2010; Cella et al., 2019) | 1 week before the intervention begins, immediately after intervention ends (approximately 7 weeks)
  Measures symptoms of anxiety

SECONDARY OUTCOMES:
Three Item Loneliness Scale (Hughes et al., 2004) | 1 week before the intervention begins, immediately after intervention ends (approximately 7 weeks)
  Measures feelings of loneliness
PROMIS Social Isolation 8a (Cella et al., 2010) | 1 week before the intervention begins, immediately after intervention ends (approximately 7 weeks)
  Measures feelings of social isolation
PROMIS Emotional Support 8a (Cella et al., 2010) | 1 week before the intervention begins, immediately after intervention ends (approximately 7 weeks)
  Measures emotional support
The Brief Measure of Mental Health Literacy Scale (Mackenzie & Reynolds, in preparation) | 1 week before the intervention begins, immediately after intervention ends (approximately 7 weeks)
  Measures mental health literacy (one's knowledge of mental health problems and services available for these mental health problems).
Demographic Information | 1 week before the intervention begins
  Gender identification, age, highest level of education completed, occupational status, marital status, living arrangement, location of residence, and racial and ethnic background.

CONTACTS AND LOCATIONS:
Overall Officials: Inga A Christianson, BA, Principal Investigator — The University of Manitoba; Kristin Reynolds, Ph.D., Principal Investigator — The University of Manitoba
Locations (1):
- The University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share this data.

REFERENCES:
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Cella D, Choi SW, Condon DM, Schalet B, Hays RD, Rothrock NE, Yount S, Cook KF, Gershon RC, Amtmann D, DeWalt DA, Pilkonis PA, Stone AA, Weinfurt K, Reeve BB. PROMIS(R) Adult Health Profiles: Efficient Short-Form Measures of Seven Health Domains. Value Health. 2019 May;22(5):537-544. doi: 10.1016/j.jval.2019.02.004. PMID 31104731
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- See also: Statistics Canada. (2019). Population Projections: Canada, provinces, and territories, 2018 to 2068. Statistics Canada. — https://www150.statcan.gc.ca/n1/en/daily-quotidien/190917/dq190917b-eng.pdf?st=uXx6TuhX